CLINICAL TRIAL: NCT00986674
Title: Three-Arm Randomized Phase II Study of Carboplatin and Paclitaxel in Combination With Cetuximab, IMC-A12 or Both in Patients With Advanced Non-Small Cell Lung Cancer Who Will Not Receive Bevacizumab-Based Therapy
Brief Title: Carboplatin and Paclitaxel Combined With Cetuximab and/or IMC-A12 in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01976; E4508 (Other: Eastern Cooperative Oncology Group); U10CA021115 (NIH)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-03

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
Keywords: Advanced Non-small Cell Lung Cancer; Carboplatin; Paclitaxel; Cetuximab; IMC-A12
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cixutumumab; Carboplatin; Paclitaxel; Taxes; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (carboplatin, paclitaxel, cetuximab) (Experimental): Patients receive carboplatin IV over 15-30 minutes and paclitaxel IV over 3 hours on days 1 and 22 and cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 42 days for 2 courses. Patients with stable or responding disease after 2 courses proceed to maintenance therapy with cetuximab alone on days 1, 8, 15, 22, 29, and 36. Treatment with cetuximab repeats every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Biological: cetuximab
- Arm II (carboplatin, paclitaxel, cixutumumab) (Experimental): Patients receive carboplatin and paclitaxel as in arm I. Patients also receive cixutumumab IV over 1 hour on days 1, 15, and 29. Treatment repeats every 42 days for 2 courses. Patients with stable or responding disease after 2 courses proceed to maintenance therapy with cixutumumab alone on days 1, 15, and 29. Treatment with cixutumumab repeats every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cixutumumab; Drug: carboplatin; Drug: paclitaxel
- Arm III (carboplatin, paclitaxel, cetuximab, cixutumumab) (Experimental): Patients receive carboplatin, paclitaxel, and cetuximab as in arm I. Patients also receive cixutumumab as in arm II. Treatment repeats every 42 days for 2 courses. Patients with stable or responding disease after 2 courses proceed to maintenance therapy with cetuximab as in arm I and cixutumumab as in arm II.
  Interventions: Biological: cixutumumab; Drug: carboplatin; Drug: paclitaxel; Biological: cetuximab

INTERVENTIONS:
Biological: cixutumumab — Given IV
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
  Arms: Arm II (carboplatin, paclitaxel, cixutumumab); Arm III (carboplatin, paclitaxel, cetuximab, cixutumumab)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
  Arms: Arm I (carboplatin, paclitaxel, cetuximab); Arm III (carboplatin, paclitaxel, cetuximab, cixutumumab)

SUMMARY:
This randomized phase II trial is studying how well giving carboplatin and paclitaxel together with cetuximab and/or cixutumumab (IMC-A12) works in treating patients with stage IIIB or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab and cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy together with monoclonal antibody therapy may kill more tumor cells. It is not yet known whether carboplatin and paclitaxel are more effective when given with cetuximab and/or cixutumumab in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression-free survival of patients with non-small cell lung cancer (NSCLC) randomized to carboplatin plus paclitaxel plus cetuximab or carboplatin plus paclitaxel plus cixutumumab (IMC-A12) or carboplatin plus paclitaxel plus cetuximab plus cixutumumab.

SECONDARY OBJECTIVES:

I. To evaluate the response rate, disease control rate (complete response plus partial response plus stable disease), and toxicities for each arm.

II. To evaluate epidermal growth factor receptor (EGFR) by Immunohistochemistry (IHC), mutation, and gene copy number, Insulin-like growth factor 1 receptor (IGF-1R) and Insulin-like growth factor 2 receptor (IGF-2R) expression (both phosphorylated and unphosphorylated states), expression of p-AKT (ie, Protein Kinase B) by IHC, and k-ras mutation.

III. Plasma-based biomarkers will be evaluated for total and free insulin-like growth factor 1 and 2, IGF-growth factor binding protein 3 (IGFBP3) and circulating levels of epidermal growth factor (EGF) and Transforming growth factor (TGF) alpha.

IV. To evaluate overall survival on each of the three arms.

OUTLINE: This is a multicenter study. Patients are stratified according to gender and histology (squamous cell vs non-squamous cell). Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive carboplatin intravenously (IV) over 15-30 minutes and paclitaxel IV over 3 hours on days 1 and 22 and cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 42 days for 2 courses. Patients with stable or responding disease after 2 courses proceed to maintenance therapy with cetuximab alone on days 1, 8, 15, 22, 29, and 36. Treatment with cetuximab repeats every 42 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive carboplatin and paclitaxel as in arm I. Patients also receive cixutumumab IV over 1 hour on days 1, 15, and 29. Treatment repeats every 42 days for 2 courses. Patients with stable or responding disease after 2 courses proceed to maintenance therapy with cixutumumab alone on days 1, 15, and 29. Treatment with cixutumumab repeats every 42 days in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive carboplatin, paclitaxel, and cetuximab as in arm I. Patients also receive cixutumumab as in arm II. Treatment repeats every 42 days for 2 courses. Patients with stable or responding disease after 2 courses proceed to maintenance therapy with cetuximab as in arm I and cixutumumab as in arm II.

Tumor tissue samples are collected at baseline for analysis of EGFR expression by IHC, mutation, and gene copy number; IGF-1R and IGF-2R expression (both phosphorylated and unphosphorylated states); p-AKT expression by IHC; and k-ras mutation. Blood, serum, and plasma samples are collected periodically for biomarker analysis.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: 200 patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB disease

    * T4, NX with nodule in ipsilateral lung lobe allowed provided patient is not a candidate for combined chemotherapy and radiotherapy
  * Stage IV disease (includes M1a and M1b)
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Ineligible for or refused treatment with bevacizumab
* No untreated or symptomatic central nervous system (CNS) metastases

  * Patients with a history of CNS metastases that are definitively treated, stable, and controlled are eligible provided the following criteria are met:

    * Definitive therapy (surgery and/or radiotherapy) has been administered
    * Not planning to undergo additional treatment for brain metastases
    * Clinically stable
    * Off corticosteroids or on a stable dose of corticosteroids for ≥ 14 days before study entry
* ECOG performance status 0-1
* Leukocytes > 3,000/mm^3
* Absolute neutrophil count (ANC) > 1,500/mm^3
* Hemoglobin > 9 g/dL
* Platelet count > 100,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate Aminotransferase (AST) < 3 times ULN (< 5 times ULN if elevations due to liver metastases)
* Creatinine < 1.5 times ULN OR creatinine clearance > 60 mL/min
* Fasting serum glucose < 120 mg/dL
* Partial thromboplastin time (PTT) ≤ 1.2 times ULN and international normalized ratio (INR) ≤ 1.5 (unless patient is on anticoagulation therapy)
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after the last dose of cixutumumab
* No poorly controlled diabetes mellitus

  * Patients with a history of diabetes mellitus are eligible provided their blood glucose is within normal range and they are on a stable dietary or therapeutic regimen for this condition
* No other prior or concurrent malignancy, except for the following:

  * Curatively treated malignancy with no known active disease for ≥ 3 years AND is considered to be at low risk for recurrence by the treating physician
  * Adequately treated nonmelanoma skin cancer or lentigo maligna with no evidence of disease
  * Adequately treated cervical carcinoma in situ with no evidence of disease
  * Prostatic intraepithelial neoplasia with no evidence of prostate cancer
* Concurrent therapeutic anticoagulation allowed provided there is no bleeding and patient is on a stable dose of anticoagulation therapy (e.g., Warfarin with an INR of 2-3) for > 2 weeks prior to study entry
* At least 21 days since prior radiotherapy
* More than 4 weeks since prior major surgery or hormonal therapy (other than hormone replacement therapy) and recovered
* More than 1 year since prior neoadjuvant or adjuvant chemotherapy

Exclusion criteria:

* Small cell lung cancer or mixed small cell and NSCLC
* History of allergic reactions attributed to compounds of similar chemical or biological composition to cixutumumab
* History of any medical or psychiatric condition, addictive disorder, or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with study participation or study treatments or may interfere with the conduct of the study or interpretation of study results
* Prior agents targeting the EGFR or Insulin-like growth factor (IGFR) pathways
* Prior therapy for advanced NSCLC, except for surgery and/or radiotherapy
* Prior systemic therapy, including bevacizumab for advanced stage NSCLC
* Pregnant or nursing
* Peripheral neuropathy > grade 1 as per Common Terminology Criteria for Adverse Event (CTCAE) v 4.0
* History of or suspected interstitial pneumonitis or pulmonary fibrosis on imaging
* Significant uncontrolled cardiac disease within the past 6 months, including any of the following:

  * Uncontrolled hypertension (BP > 150/100 mm Hg)
  * Unstable angina
  * Recent myocardial infarction
  * Uncontrolled congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* Arterial thrombosis, pulmonary embolus, deep vein thrombosis, or hemorrhagic disorders within the past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, Principal Investigator — Indiana University School of Medicine
Locations (249):
- United States (249):
  - Stanford University Hospitals and Clinics, Stanford, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Medical Center of Central Georgia, Macon, Georgia
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett, Lafayette, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium CCOP, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - New York Oncology Hematology PC - Latham, Latham, New York
  - New York Oncology Hematology PC - Rexford, Rexford, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - West Virginia University Charleston, Charleston, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - UW Health Oncology - 1 South Park, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on September 11, 2009. The trial was suspended to accrual on December 17, 2010 after accruing 140 patients and accrual was subsequently terminated on April 19, 2011 due to excessive grade 5 events within 30 days of study registration.
Period: Overall Study
Arm/Group | Arm I (Carboplatin, Paclitaxel, Cetuximab) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab)
Started | 47 | 45 | 48
Treated | 43 | 42 | 47
Eligible and Treated | 39 | 41 | 47
Completed | 0 | 0 | 0
Not Completed | 47 | 45 | 48
Not completed — Lack of Efficacy | 28 | 25 | 23
Not completed — Adverse Event | 4 | 8 | 9
Not completed — Death | 5 | 0 | 4
Not completed — Withdrawal by Subject | 6 | 2 | 1
Not completed — alternative therapy | 0 | 0 | 1
Not completed — not start protocol therapy | 4 | 3 | 1
Not completed — unknown/not specify | 0 | 7 | 9

BASELINE CHARACTERISTICS:
Population: The primary population is eligible and treated patients in the study. Both baseline analysis and efficacy outcomes are based on this primary population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Carboplatin, Paclitaxel, Cetuximab) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab) | Total
Number analyzed (Participants) | 39 | 41 | 47 | 127
Age, Continuous [Median (Full Range); unit: years] | 60 [42 to 89] | 60 [43 to 81] | 60 [44 to 76] | 60 [42 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 22 | 58
  Male | 20 | 24 | 25 | 69

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival is defined as time from registration to disease progression or death from any cause, whichever occurred earlier. Disease progression was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions .
  All eligible and treated patients were included in the analysis.
Time Frame: Tumor measurements are repeated every 6 weeks while on treatment. After off treatment, assessed every 3 months if patient is < 2 years from study entry and every 6 months in year 3
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Carboplatin, Paclitaxel, Cetuximab) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab)
Number analyzed (Participants) | 39 | 41 | 47
months | 3.4 [2.6 to 5.8] | 4.2 [3.5 to 5.3] | 4.0 [3.2 to 5.4]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from registration to death from any cause.
Time Frame: assessed every 3 months if patient is < 2 years from study entry and every 6 months in year 3
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Carboplatin, Paclitaxel, Cetuximab) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab)
Number analyzed (Participants) | 39 | 41 | 47
months | 9.8 [7.4 to 17.2] | 7.7 [5.8 to 11.5] | 8.8 [7.2 to 14.9]

3. Secondary Outcome: Response Rate
Description: Tumor response was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Complete response (CR) was defined disappearance of all tumor lesions. Partial response (PR) was defined as as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter. Overall response rate= CR+PR.
Time Frame: as for outcome 1
Population: eligible and treated patients who have response data. 3 patients on arm I and 1 patient on arm III had unknown/missing tumor response and were excluded from the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Carboplatin, Paclitaxel, Cetuximab) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab)
Number analyzed (Participants) | 36 | 41 | 46
percentage of participants | 11.1 [3.1 to 26.1] | 22.0 [10.6 to 37.6] | 21.7 [10.9 to 36.4]

ADVERSE EVENTS:
Time Frame: Assessed every cycle (6 weeks) while on treatment and for 30 days after the end of treatment.
Description: After off treatment, patients were assessed every 3 months if <2 years and every 6 months in year 3 to report any reportable long-term toxicity occurring prior to diagnosis of progression/relapse that has not been previously reported.
Arm/Group | Arm I (Carboplatin, Paclitaxel, Cetuximab) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab)
Serious Adverse Events (participants affected / at risk) | 27/44 | 27/42 | 36/48
Other Adverse Events (participants affected / at risk) | 43/44 | 40/42 | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Carboplatin, Paclitaxel, Cetuximab) (N=44) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) (N=42) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab) (N=48)
Anemia (Blood and lymphatic system disorders) | 6 | 3 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Edema face (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 7 | 5
Pain (General disorders) | 0 | 0 | 1
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 3
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 4
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2
Allergic reaction (Immune system disorders) | 0 | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 0 | 1
Bladder infection (Infections and infestations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 4 | 0 | 1
Lymph gland infection (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 2 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 2
Neutrophil count decreased (Investigations) | 12 | 13 | 20
Platelet count decreased (Investigations) | 3 | 5 | 4
Urine output decreased (Investigations) | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 8 | 6 | 8
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Carboplatin, Paclitaxel, Cetuximab) (N=44) | Arm II (Carboplatin, Paclitaxel, Cixutumumab) (N=42) | Arm III (Carboplatin, Paclitaxel, Cetuximab, Cixutumumab) (N=48)
Anemia (Blood and lymphatic system disorders) | 29 | 28 | 29
Chills (General disorders) | 3 | 7 | 7
Edema limbs (General disorders) | 4 | 0 | 0
Fatigue (General disorders) | 31 | 30 | 37
Fever (General disorders) | 4 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 22 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 5 | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 2 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 6 | 13
Rash acneiform (Skin and subcutaneous tissue disorders) | 30 | 6 | 29
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 3 | 11
Constipation (Gastrointestinal disorders) | 9 | 10 | 8
Diarrhea (Gastrointestinal disorders) | 17 | 15 | 19
Dyspepsia (Gastrointestinal disorders) | 5 | 4 | 4
Mucositis oral (Gastrointestinal disorders) | 16 | 11 | 21
Nausea (Gastrointestinal disorders) | 20 | 27 | 20
Vomiting (Gastrointestinal disorders) | 10 | 14 | 13
Alanine aminotransferase increased (Investigations) | 7 | 2 | 4
Alkaline phosphatase increased (Investigations) | 6 | 5 | 6
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 4
Cholesterol high (Investigations) | 0 | 5 | 7
Creatinine increased (Investigations) | 0 | 5 | 2
Lipase increased (Investigations) | 0 | 3 | 1
Lymphocyte count decreased (Investigations) | 4 | 0 | 5
Neutrophil count decreased (Investigations) | 9 | 12 | 6
Platelet count decreased (Investigations) | 13 | 14 | 19
Serum amylase increased (Investigations) | 3 | 2 | 2
Weight loss (Investigations) | 12 | 15 | 19
White blood cell decreased (Investigations) | 10 | 10 | 10
Investigations - Other, specify (Investigations) | 0 | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 17 | 23 | 25
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 4
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 7 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 16 | 11
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 9 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 5 | 5
Hypokalemia (Metabolism and nutrition disorders) | 7 | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 13 | 7 | 17
Hyponatremia (Metabolism and nutrition disorders) | 5 | 9 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 13 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 12 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3
Dizziness (Nervous system disorders) | 3 | 6 | 5
Dysgeusia (Nervous system disorders) | 8 | 7 | 8
Headache (Nervous system disorders) | 6 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 19 | 20 | 18
Flashing lights (Eye disorders) | 0 | 3 | 1
Floaters (Eye disorders) | 0 | 5 | 1
Insomnia (Psychiatric disorders) | 3 | 1 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Hematuria (Renal and urinary disorders) | 1 | 0 | 3
Hypotension (Vascular disorders) | 1 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less